CLINICAL TRIAL: NCT06989905
Title: Operant Conditioning of the Wrist Extensor Motor Evoked Potential to Target Corticospinal Plasticity and Upper Limb Motor Recovery After Cervical Spinal Cord Injury
Brief Title: MEP Up-conditioning to Target Corticospinal Plasticity
Acronym: uMEP2
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Doscher Neurorehabilitation Research Program (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Allison Lewis, Post-doctoral Scholar, Principal Investigator, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00138869; 1K99HD117041 (NIH)
Record Dates: First submitted 2025-05-08; First posted 2025-05-25 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injury; Tetraplegia/Tetraparesis
Keywords: Central Nervous System; Nervous System; Rehabilitation Studies; Spinal Cord; spinal cord injury; upper extremity; upper limb; motor impairment; tetraplegia; quadriplegia
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia; Neurologic Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Operant Up-Conditioning of the Motor Evoked Potential (Experimental): The intervention consists of approximately 6 baseline sessions and 24 conditioning sessions at a pace of 3 sessions/week, 1-2 hour duration, over 10 weeks. At the beginning of each session, electromyographic (EMG) recording and nerve stimulating electrodes are placed over the arm. In all sessions, motor evoked potentials (MEPs) will be measured while the sitting subject provides a pre-set level of background muscle EMG with joint angles fixed. In 225 control trials of each baseline sessions and the first 20 trials of conditioning sessions the subject will receive no feedback as to MEP size (i.e., control MEPs). In 225 conditioning trials of each conditioning session, the subject will be encouraged to increase the target muscle MEP, and will receive immediate feedback as to whether MEP size was above a criterion (i.e., whether the trial was a success).
  Interventions: Behavioral: Up-conditioning of the wrist extensor motor evoked potential

INTERVENTIONS:
Behavioral: Up-conditioning of the wrist extensor motor evoked potential — At the beginning of each session, EMG recording and nerve stimulating electrodes are placed over the arm. In all sessions, MEPs will be measured while the sitting subject provides a pre-set level of background muscle EMG with joint angles fixed. In 225 control trials of each baseline sessions and the first 20 trials of conditioning sessions the subject will receive no feedback as to MEP size (i.e., control MEPs). In 225 conditioning trials of each conditioning session, the subject will be encouraged to increase the target muscle MEP, and will receive immediate feedback as to whether MEP size was above a criterion (i.e., whether the trial was a success).

SUMMARY:
Individuals with chronic cervical spinal cord injury will complete a 10-week training protocol where participants receive non-invasive brain stimulation and feedback on the size of the corresponding muscle response (wrist extensor).

Investigators will assess the impact of the brain stimulation training on 1) the brain-to-spinal cord-to-muscle connection and 2) motor functions of the arm and hand. Also, brain and spine magnetic resonance imaging will be collected before and after the training. The imaging measurements will tell investigators about how spinal damage, brain function, and brain structure relate to motor presentation and the response to the training.

DETAILED DESCRIPTION:
Corticospinal function is essential in generating and controlling voluntary movements. Cervical spinal cord injury (SCI) disrupts corticospinal connections, therefore, often results in weak voluntary activation of muscles and impaired motor control in the upper limb (UL). An intervention that improves corticospinal function could enhance motor function recovery; however, such interventions are not currently readily available to people with incomplete SCI. Operant up-conditioning of a motor evoked potential (MEP) to transcranial magnetic stimulation (non- invasive brain stimulation) that can increase corticospinal excitability for the targeted muscle may be able to fill this gap. The overarching hypothesis is that targeting beneficial plasticity to the corticospinal pathway can change the brain and spinal cord and improve upper limb motor function in people with chronic cervical SCI. As initial steps towards testing this, the proposed project aims to apply MEP operant up-conditioning in the wrist extensor of the affected UL, improve corticospinal activation of the wrist extensor, and thereby improve motor functions in which the wrist is involved in individuals with cervical SCI. Recent studies suggest that MEP up- conditioning is feasible and can increase MEP size that reflects corticospinal excitability. Building on those studies, this project will examine the effects of wrist extensor MEP operant up-conditioning in people with chronic cervical SCI. Individuals with weak wrist extension due to incomplete cervical SCI will undergo a standard MEP up-conditioning protocol (6 baseline and 24 up-conditioning sessions over 10 weeks). Before and after the intervention period, neurophysiological measurements, clinical and functional assessments, neuroimaging of the spinal cord and brain will be performed. The results will facilitate development and clinical translation of MEP operant conditioning as a novel non-invasive therapy that may complement other therapies and further enhance motor function recovery in people with SCI or other disorders.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 yrs old)
* A history of injury to spinal cord at or above C6
* >6 months post SCI
* Weak wrist extension at least unilaterally
* Expectation that current medication will be maintained without change for at least 3 months. Stable use of anti-spasticity medication (e.g., baclofen, diazepam, tizanidine) is accepted.

Exclusion Criteria:

* Motoneuron injury
* Medically unstable condition
* Cognitive impairment
* A history of epileptic seizures
* Metal implants in the cranium
* Implanted biomedical device in or above the chest (e.g., a cardiac pacemaker, cochlear implant)
* Extensive use of functional electrical stimulation to the arm on a daily basis
* Pregnancy (due to changes in posture and potential medical instability)
* Contraindications to MRI
* No measurable MEP elicited in the ECR
* Unable to produce any voluntary ECR EMG activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Extensor Carpi Radialis (ECR) Motor Evoked Potential (MEP) amplitude | Reported as an average of the 6 baseline sessions (over weeks 1-2) and average of the last 6 conditioning sessions (over weeks 8-10)
  Size of MEP elicited at the fixed stimulus intensity (e.g., ~ 10-15% maximum stimulator output) of transcranial magnetic stimulation (TMS) above motor threshold) (in %M wave maximum amplitude)

SECONDARY OUTCOMES:
Maximum Voluntary Contraction - ECR | Reported as an average of the 6 baseline sessions (over weeks 1-2) and average of the last 6 conditioning sessions (over weeks 8-10)
  Maximum voluntary contraction measured by electromyography (EMG) (in mV); average of two trials
Capabilities Upper Extremity Test (CUE-T) | Baseline, after the 24th conditioning session (typically within 1 week), 1 month and 3 months post
  The CUE-T is an objective clinical measure of a person with tetraplegia's ability to complete actions with the arm and hand. This scale measures motor function. It consists of 19 tasks (17 unilateral, 2 bilateral). Scoring is based completion of the action, number of repetitions, or time to complete depending on the item and converted from raw score to 5-point scale (0-4, 4 is best).
Graded and Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP) | Baseline, after the 24th conditioning session (typically within 1 week), 1 month and 3 months post
  The GRASSP is a clinical impairment measure to assess sensorimotor hand function in people with cervical SCI. The GRASSP tests 3 domains of hand function including strength, sensibility, and prehension. The GRASSP contains 6 tasks for each side scored from 0-5 for a possible score of 0-30 per side or 0-60 total, where higher scores are better.
Spinal Cord Independence Measure (SCIM III) | Baseline, after the 24th conditioning session (typically within 1 week), 1 month and 3 months post
  The SCIM is a self-report survey of daily activity independence in self-care, respiration and sphincter management, and mobility. The scores range from 0-100, where higher scores represent greater independence.
Life Situation Questionnaire Revised (LSQ-R) | Baseline, after the 24th conditioning session (typically within 1 week), 1 month and 3 months post
  The LSQ-R is a self-report survey of quality of life that contains 20 life satisfaction items and 30 life problems items. All items are evaluated using a 5-point scale. For the satisfaction items, a score of 1 indicates "very dissatisfied," while a score of 5 denotes "very satisfied." For the problems items, a score of 1 represents "no problem," and a score of 5 signifies a "major problem."

OTHER OUTCOMES:
ECR MEP recruitment curve | Baseline, after the 24th conditioning session (typically within 1 week), 1 month and 3 months post
  Maximum MEP size (in mV and %maximum M-wave (Mmax)) and active MEP threshold (in %maximum stimulator output (MSO)
Silent Period Duration | Reported as an average of the 6 baseline sessions (over weeks 1-2) and average of the last 6 conditioning sessions (over weeks 8-10)
  Silent period duration measured as the time from the start of the MEP to the recovery of EMG activity to the prestimulus level (ms)
Spine imaging - lesion overlap with lateral corticospinal tract (LCST) or motor tract damage | Baseline
  Percent by volume of overlap between lesion and the LCST
Spine imaging - Lesion volume | Baseline
  Volume of the lesion from the lesion segmentation in cubic millimeters
Brain imaging - Diffusion Kurtosis Imaging (DKI) - Kurtosis Fractional Anisotropy | Baseline
  Kurtosis fractional anisotropy (KFA) is a ratio value that reflects the directional variation of non-Gaussian water diffusion, reflecting tissue complexity.
Brain Imaging - Diffusion Kurtosis Imaging - Axial Kurtosis | Baseline
  Axial kurtosis (AK) is the kurtosis along the axial direction of the diffusion ellipsoid; closer to 0 in white matter, because it represents less diffusion restriction.
Brain imaging - Resting state connectivity of sensorimotor network | Baseline
  Connectivity between pairs of brain regions as Fisher's z transformed correlation coefficients. Brain regions in the sensorimotor network include primary motor cortex (M1), somatosensory cortex (S1), ventral premotor (PMv), dorsal premotor (PMd), supplementary motor area (SMA), and pre-supplementary motor area (preSMA).
Brain Imaging - Diffusion Tensor - Fractional Anisotropy | Baseline
  Corticospinal tract fractional anisotropy (FA) measures general microstructural integrity.
  FA is a ratio value where values closer to 1 suggest greater anisotropy of water diffusion, suggesting a tendency for water to diffuse in a single direction and greater structural integrity.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Lewis, DPT, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with the OpenNEURO repository (MRI data) and the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Data and Specimen Hub (DASH) (clinical assessments and EMG data).
Access Criteria: Data on NICHD DASH is available via controlled access. The requester must provide details about the study, funding source, principal investigator, and the names and email addresses of the authorized representative or Institutional Business Official, as well as any affiliated personnel. Additionally, the submission must include the NICHD DASH Data Use Agreement and, if required by the requested study, IRB Approval for Data Request. The requesting institution must also maintain active Federalwide Assurance (FWA) status
  MRI data in OpenNEURO is open to the public. Participants can opt in or out of sharing MRI data.